CLINICAL TRIAL: NCT07132099
Title: RCT Comparing ASSIP and ACT on Mental Pain and Suicidal Ideation in Individuals With Suicide Attempts
Brief Title: Randomized Suicide Prevention Trial Using ASSIP and ACT in Suicide Attempters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ardakan University (Other)
Responsible Party: Principal Investigator, Hadiseh Yaghoobi, Researcher, Master of General Psychology Student, Ardakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.ARDAKAN.REC.1404.002
Record Dates: First submitted 2025-08-11; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Suicide; Suicide Ideation
Keywords: Attempted Suicide Short Intervention Program; Acceptance and Commitment Therapy; Suicidal Ideation; Mental Pain; Suicide attempt; ASSIP; ACT
MeSH Terms: conditions — Suicide; Suicidal Ideation; Suicide, Attempted | interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with three parallel groups. Participants will be randomly assigned to one of these three groups. The first group will receive ASSIP alongside treatment as usual (TAU) , the second group will receive ACT alongside TAU , and the third group (the control group) will receive only TAU. All groups will receive their interventions simultaneously and in parallel for the duration of the study.
Who Masked: Participant
Masking Description: Only participants will be unaware of their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASSIP + TAU (Experimental): Participants in this group receive the Attempted Suicide Short Intervention Program (ASSIP) in addition to treatment as usual (TAU).
  Interventions: Behavioral: Attempted Suicide Short Intervention Program (ASSIP); Other: Treatment as Usual (TAU)
- ACT + TAU (Experimental): Participants in this group receive Acceptance and Commitment Therapy (ACT) alongside treatment as usual (TAU).
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Other: Treatment as Usual (TAU)
- Control Group (TAU only) (Other): This control group receives only treatment as usual (TAU).
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Attempted Suicide Short Intervention Program (ASSIP) — This is a brief, structured, patient-centered therapy consisting of three to four face-to-face sessions. Each session typically lasts between 60 to 90 minutes. A fourth session may be added if clinically necessary.
  Arms: ASSIP + TAU
Behavioral: Acceptance and Commitment Therapy (ACT) — This intervention uses the "ACT for Life" protocol, which is designed to maximize recovery after suicidal crises. It consists of three components delivered over three to six individual sessions. The average number of sessions is four to five, with each session lasting approximately 60 minutes.
  Arms: ACT + TAU
Other: Treatment as Usual (TAU) — Treatment as usual (TAU) is not a structured intervention within this study. It may include standard outpatient or inpatient services, pharmacotherapy, or no structured treatment, depending on individual circumstances.

SUMMARY:
This is a randomized controlled trial that aims to compare the effectiveness of two psychological treatment approaches: the Attempted Suicide Short Intervention Program (ASSIP) and Acceptance and Commitment Therapy (ACT). The study seeks to determine which of these two methods is more effective in reducing suicidal ideation and mental pain in individuals who have recently attempted suicide.

In this study, 60 participants with a history of suicide attempts will be randomly assigned to three groups. One group will receive ASSIP in addition to treatment as usual (TAU), the second group will receive ACT alongside TAU, and the third group will be a control group receiving TAU only. The results will be assessed using the Beck Scale for Suicide Ideation (BSSI) and the Orbach & Mikulincer Mental Pain Scale (OMMP) at three stages: pre-test, post-test, and follow-up.

The ultimate goal of this research is to provide valuable insights into the comparative effectiveness of ASSIP and ACT interventions for suicide attempters and to contribute to evidence-based suicide prevention strategies. The findings are expected to inform clinical practice and guide future research in this field.

DETAILED DESCRIPTION:
Background and Rationale:

Suicide attempts are a major global public health concern and one of the leading causes of premature mortality, particularly among individuals aged 15 to 29 years. In Iran, as in many countries, suicide attempts represent a critical mental health issue requiring effective, evidence-based interventions. Two therapeutic approaches have demonstrated promising results in reducing suicidal ideation and preventing repeated attempts: the Attempted Suicide Short Intervention Program (ASSIP) and Acceptance and Commitment Therapy (ACT).

ASSIP is a brief, structured, narrative-based intervention developed to address the underlying personal crisis and cognitive-behavioral mechanisms that lead to suicidal behavior. It typically involves three to four sessions, followed by long-term follow-up contacts. ACT is a third-wave behavioral therapy aimed at increasing psychological flexibility and reducing experiential avoidance, often associated with suicidal crises.

Despite evidence supporting both methods internationally, little research has compared their effectiveness in the Iranian context.

Study Overview:

This randomized controlled trial will enroll 60 adults with a recent history of suicide attempt, identified through the Eslamshahr Health Network. Participants will be randomly assigned to one of three groups:

1. ASSIP plus treatment as usual (TAU)
2. ACT plus TAU
3. TAU only (control) Interventions will be delivered in an outpatient health center setting. The ASSIP group will receive three core sessions (with a possible fourth session) delivered according to the official ASSIP manual. The ACT group will receive four to five individual sessions following the "ACT for Life" protocol, specifically adapted for suicide prevention.

Assessment and Follow-up:

The primary outcomes are suicidal ideation and mental pain, assessed using validated Persian versions of the Beck Scale for Suicide Ideation (BSSI) and the Orbach & Mikulincer Mental Pain Scale (OMMP). Assessments will occur at baseline (pre-test), immediately after treatment (post-test), and one month after intervention (follow-up). Data will be analyzed using SPSS v27, applying descriptive statistics, analysis of covariance, and post hoc comparisons.

Significance:

This study is expected to generate context-specific evidence on the comparative effectiveness of ASSIP and ACT in reducing suicidal ideation and mental (or psychological) pain in Iranian suicide attempters. The findings will help inform mental health services in Iran and contribute to global suicide prevention strategies by clarifying which short-term, evidence-based intervention is more effective and feasible in similar healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Having the ability to read and write
* Providing informed consent to participate in the study
* Having at least one suicide attempt in the past 4 months

Exclusion Criteria:

* Having a severe psychiatric or physical illness that interferes with the treatment process
* Receiving concurrent structured psychological interventions (other than TAU) that may interfere with the study's treatment process.
* Lack of informed consent to participate in the study
* Substance abuse based on DSM-5 criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mental Pain | pre-intervention, immediately following the intervention, and at 1-month follow-up
  This measure assesses the intensity of mental pain using the 44-item Orbach & Mikulincer Mental Pain Scale (OMMP). The scale has nine subscales to measure various aspects of mental pain, including inevitability, lack of control, narcissism/worthlessness, emotional turmoil, numbness, alienation, confusion, social withdrawal, and emptiness (meaninglessness).
Suicidal Ideation | pre-intervention, immediately following the intervention, and at 1-month follow-up
  This measure assesses suicidal thoughts, attitudes, and behaviors using the 19-item self-report Beck Scale for Suicide Ideation (BSSI). Each item is rated on a Likert scale from 0 to 2, with a total score ranging from 0 to 38. A score of 0-5 indicates no suicidal ideation, 6-19 suggests the presence of suicidal thoughts, and 20-38 signifies a high level of suicide ideation and planning.

CONTACTS AND LOCATIONS:
Overall Officials: Azadeh Choobforoushzadeh, PhD, Study Director — Ardakan University; Marjan Fathi, Postdoctoral, Study Director — Iran University of Medical Sciences
Locations (1):
- The Imam Hossein District Health Center, Eslamshahr, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to the highly sensitive and confidential nature of the data collected from suicide attempters. The protocol for this study will be published in a scientific journal upon peer review approval. Furthermore, after data collection and analysis are complete, the results will be published in a scientific journal following peer review approval.

REFERENCES:
- [Background] Olfson M, Wall M, Wang S, Crystal S, Liu SM, Gerhard T, Blanco C. Short-term Suicide Risk After Psychiatric Hospital Discharge. JAMA Psychiatry. 2016 Nov 1;73(11):1119-1126. doi: 10.1001/jamapsychiatry.2016.2035. PMID 27654151
- [Background] World Health Organization. (2025). Suicide. https://www.who.int/news-room/fact-sheets/detail/suicide
- [Background] Shneidman ES. The psychological pain assessment scale. Suicide Life Threat Behav. 1999 Winter;29(4):287-94. No abstract available. PMID 10636323
- [Background] Shirani Isfahani, N., Mohammadpanah Ardakan, A., & Rezapoor Mirsaaleh, M. (2023). Lived emotional experiences of women who attempt suicide. Journal of Health System Research, 19(4), 325-335. (in Persian)
- [Background] Pompili M. On mental pain and suicide risk in modern psychiatry. Ann Gen Psychiatry. 2024 Jan 16;23(1):6. doi: 10.1186/s12991-024-00490-5. PMID 38229110
- [Background] Mojahedi M, Esmaeili A, Mahdizadeh K, Nakhaei MH, Salehiniya H, Sahranavard S. Trends of suicide attempts and factors related to completed suicide during the years 2014-2019 in South Khorasan province, Iran. Asian J Psychiatr. 2021 Nov;65:102825. doi: 10.1016/j.ajp.2021.102825. Epub 2021 Sep 2. PMID 34562752
- [Background] Karami, J., Begian Kuleh Marz, M. J., Momeni, Kh., & Elahi, A. (2018). Measurement of psychological pain: Psychometric properties and confirmatory factor analysis of the One-Dimensional Multidimensional Pain Questionnaire (OMMP). Health Psychology, 7(25), 146-172. (in Persian)
- [Background] Hosseini, A., Jamshidi, T., Sedghi, S., Jalali, M., & Shamsi, F. (2019). Effectiveness of a suicide prevention training program based on SOS in reducing suicidal ideation and depression in girls. Journal of Nursing and Midwifery, 17(3), 192-203. (in Persian)
- [Background] Rizvi A, Harmer B, Saadabadi A. Suicidal Ideation. 2024 Apr 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK565877/ PMID 33351435
- [Background] Gysin-Maillart A, Schwab S, Soravia L, Megert M, Michel K. A Novel Brief Therapy for Patients Who Attempt Suicide: A 24-months Follow-Up Randomized Controlled Study of the Attempted Suicide Short Intervention Program (ASSIP). PLoS Med. 2016 Mar 1;13(3):e1001968. doi: 10.1371/journal.pmed.1001968. eCollection 2016 Mar. PMID 26930055
- [Background] Feyzollahi S, Narimany M, Mosazadeh T. (2021). Effectiveness of Acceptance and Commitment Therapy on Suicidal Thoughts, Self-concealment and Cognitive Emotion Regulation in Women with Suicidal Thoughts. Rooyesh. 10(2), 69-80. (in Persian)
- [Background] Favril L, Yu R, Geddes JR, Fazel S. Individual-level risk factors for suicide mortality in the general population: an umbrella review. Lancet Public Health. 2023 Nov;8(11):e868-e877. doi: 10.1016/S2468-2667(23)00207-4. PMID 37898519
- [Background] Chung DT, Ryan CJ, Hadzi-Pavlovic D, Singh SP, Stanton C, Large MM. Suicide Rates After Discharge From Psychiatric Facilities: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2017 Jul 1;74(7):694-702. doi: 10.1001/jamapsychiatry.2017.1044. PMID 28564699
- [Background] Chun HS, Michel K, Lee KU. A Case of Suicide Attempt Treated With Attempted Suicide Short Intervention Program. Psychiatry Investig. 2024 Feb;21(2):216-217. doi: 10.30773/pi.2023.0279. Epub 2024 Jan 24. No abstract available. PMID 38258293
- [Background] Charvet C, Boutron I, Morvan Y, Le Berre C, Touboul S, Gaillard R, Fried E, Chevance A. How to measure mental pain: a systematic review assessing measures of mental pain. Evid Based Ment Health. 2022 Nov;25(4):e4. doi: 10.1136/ebmental-2021-300350. Epub 2022 Jul 28. PMID 35902215
- [Background] Cassell EJ. Diagnosing suffering: a perspective. Ann Intern Med. 1999 Oct 5;131(7):531-4. doi: 10.7326/0003-4819-131-7-199910050-00009. PMID 10507963
- [Background] Barnes, S. M., Smith, G. P., Monteith, L. L., Gerber, H. R., & Bahraini, N. H. (2017). ACT for Life: Using Acceptance and Commitment Therapy to Understand and Prevent Suicide. In U. Kumar (Ed.), Handbook of Suicidal Behaviour, 485-504.
- [Background] Barnes, S. M., Borges, L. M., Smith, G. P., Walser, R. D., Forster, J. E., & Bahraini, N. H. (2021). Acceptance and commitment therapy to promote recovery from suicidal crises: A randomized controlled acceptability and feasibility trial of ACT for life. Journal of Contextual Behavioral Science, 20, 35-45.
- [Background] Alamdarian, H., Ibrahimi, M., Hadad, A., & Ghasemi, A. (2023). Predicting suicidal tendencies based on self-compassion and psychological flexibility in married women with multiple sclerosis. Journal of Sabzevar University of Medical Sciences, 30(3), 311-301. (in Persian)
- [Background] ASSIP. (n.d.). Attempted Suicide Short Intervention Program. http://www.assip.ch/
- See also: Official website of the Attempted Suicide Short Intervention Program (ASSIP). This website provides general information and background on the ASSIP protocol used in this study. — http://www.assip.ch/
- See also: Official website of the World Health Organization (WHO) with information and facts about suicide. This resource provides background statistics and data on suicide, which are referenced in the study's protocol. — https://www.who.int/news-room/fact-sheets/detail/suicide